CLINICAL TRIAL: NCT00725088
Title: Study of Rehabilitation Therapy on Patients After Acute Myocardial Infarction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ministry of Science and Technology of the People´s Republic of China (Other Government)
Responsible Party: Yong Huo, Peking University First Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2006BAI01A02-10
Record Dates: First submitted 2008-07-28; First posted 2008-07-30 (Estimated); Last update posted 2008-08-25 (Estimated); Status verified 2008-07

CONDITIONS: Acute Myocardial Infarction
Keywords: ST-Elevated Myocardial Infarction; Exercise Training; Rehabilitation
MeSH Terms: conditions — ST Elevation Myocardial Infarction | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): exercise training group
  Interventions: Behavioral: Exercise training
- 2 (No Intervention): control group

INTERVENTIONS:
Behavioral: Exercise training — Exercise training
  Arms: 1

SUMMARY:
The purpose of this study is to determine whether exercise rehabilitation can reduce mortality, reinfarction or heart failure of patients after acute myocardial infarction.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of ST-elevated myocardial infarction
* Heart function class I-II(killip classification)
* Agree to take cardiopulmonary exercise testing before discharge
* Signature of the informed consent document

Exclusion Criteria:

* History of myocardial infarction
* Acute myocardial infarction with severe complications(such as pulmonary edema, severe cardiac arrhythmia or cardiogenic shock)
* Atrial fibrillation
* Other severe diseases, such as HIV infection, malignant tumor or chronic diseases of liver, kidney or pulmonary
* Not be capable of exercise training

Ages: 35 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2006-12; Primary Completion 2008-12 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
Cardiac mortality | one year

SECONDARY OUTCOMES:
Non-fatal reinfarction, revascularization(PCI/CABG), ischemic stroke, unstable angina pectoris needs for hospitalization, severe heart failure needs for hospitalization | one year

CONTACTS AND LOCATIONS:
Overall Officials: Wei Gao, MD, Principal Investigator — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China